CLINICAL TRIAL: NCT00965315
Title: A Multicenter, Randomized, Parallel-group Study to Investigate the Efficacy of a Combination of Rosuvastatin and Fenofibrate in the Patients With Diabetes or Atherosclerotic Vascular Diseases With Metabolic Syndrome
Brief Title: A Multicenter Randomized Parallel-group Study to Investigate the Efficacy of a Combination of Rosuvastatin and Fenofibrate in the Patients With Diabetes or Atherosclerotic Vascular Diseases With Metabolic Syndrome
Status: Available | Type: Expanded Access
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200711014M
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes; CVD
Keywords: CV (cardiovascular); MI (myocardial infarction); fenofibrate; rosuvastatin; this trial is to test the hypothesis that the addition of fenofibrate on rosuvastatin would provide a further reduction in the time
MeSH Terms: conditions — Diabetes Mellitus; Myocardial Infarction

INTERVENTIONS:
Drug: Rosuvastatin,SFC fenofibrate — 1. Rosuvastatin 10 mg once daily
  2. Rosuvastatin 5 mg + SFC fenofibrate 160 mg

SUMMARY:
Diabetic patients have an excess risk of mortality due to cardiovascular diseases (CVD) compared to non-diabetics. Cardiovascular disease mortality rate is reportedly on the rise in several countries in the region, including urban China, Malaysia, Korea and Taiwan. Cardiovascular diseases and stroke are always the number 2 and 3 killers for Taiwanese population in recent years, and they really cost much from our medical resource. For treating dyslipidemia, one of the major risk factor for CVD, statins have been well documented to reduce CV deaths both for primary and secondary prevention in several large-scale trials. It has been reported that the clinical benefits of treating dyslipidemia in patients with diabetes mellitus should be at least equivalent to the benefits observed among those with cardiovascular disease. A meta-analysis of seven trials of statins found that treatment for about 5 years resulted in a 25% reduction in the combined outcome of coronary heart disease death and non-fatal myocardial infarction. Fibrates are another group of hypolipidemic drugs that regulate lipid metabolism and are used quite often in daily practice for diabetic dyslipidemia, because of its beneficial effect to reduce high TG and increase low HDL-C, which are the characteristic lipid abnormalities commonly seen in the patients with diabetes or metabolic syndrome. However, in recently published FIELD study, fenofibrate did not significantly reduce the risk of the primary outcome of coronary events in 9,795 participants with type 2 diabetes mellitus. The higher rate of starting statin therapy in patients allocated placebo might have masked a moderately larger treatment benefit. Furthermore, all the treatment trials to back up the lipid treatment guideline were conducted in Caucasians and no data about the combination therapy with fibrate and statin was published before.

ELIGIBILITY:
* Men or women aged 20-79 years
* with definite DM or atherosclerotic vascular diseases with metabolic syndrome (defined as the presence of three or more of the following risk factors:

  * abdominal obesity [waist circumference > 90 cm in men or > 80 cm in women],
* triglycerides > 150 mg/dL, HDL-cholesterol < 40 mg/dL in men or < 50 mg/dL in women, blood pressure > 130/85 mm Hg,
* or fasting glucose > 100 mg/dL) and who are qualified for lipid lowering therapy according to the Taiwanese national guidelines (LDL-C 130-190 mg/dL or TG 200-500 mg/dL with HDL-C < 40 mg/dL or TC/HDL-C > 5) will be eligible. The main exclusion criteria will be any known contraindications to statin or fibrate therapy,
* previous intolerance to statin or fibrate in low or high doses,
* liver enzyme levels more than 3 times the upper limit of normal,
* pregnancy or breastfeeding,
* nephrotic syndrome,
* uncontrolled diabetes mellitus (HbA1c > 9),
* uncontrolled hypothyroidism,
* plasma LDL-C level higher than 190 mg/dL or triglyceride level higher than 500 mg/dL,
* coronary heart disease event or revascularisation within a month, congestive heart failure (New York Heart Association classification IIIb or IV),
* hemodynamically important valvular heart disease, gastrointestinal conditions affecting absorption of drugs,
* treatment with other drugs that seriously affect the pharmacokinetics of statins or fibrate,
* unexplained creatine phosphokinase concentrations six or more times the upper limit of normal,
* life-threatening malignancy,
* treatment with immuno suppressive or other lipid lowering drugs.
* Patients previously treated with monotherapy with statins or fibrates will be qualified if they have not already had titration to a dose higher than the equivalent of 5 mg/d of rosuvastatin or 80 mg/d of SFC fenofibrate.

Ages: 20 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult